CLINICAL TRIAL: NCT01648504
Title: Integration of an Electronic Education System Into Colonoscopy: Improving Education, Consent and Compliance of Patients at Colonoscopy With an Ipad-based Secure Video Intervention
Brief Title: Johns Hopkins Interactive eGuide to Colonoscopy and Ipad Office Education to Improve Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Krames Staywell Corporation (Unknown)
Responsible Party: Principal Investigator, Ellen Stein, MD, Principal Investigator, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NA_00070166
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Colon Cancer Screening; Colon Cancer Surveillance
Keywords: Colonoscopy; Screening colonoscopy; Electronic education; Ipad; Patient education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention with eGuide to colonoscopy (Experimental): The investigators will prospectively enroll and follow patients who receive the eGuide to Colonoscopy and determine benefit and satisfaction with the intervention as part of a pilot study.
  Interventions: Other: eGuide to Colonoscopy and in office ipad education

INTERVENTIONS:
Other: eGuide to Colonoscopy and in office ipad education — The investigators will follow patients who receive in office Ipad video education and at home web portal access to the Johns Hopkins eGuide to Colonoscopy.
  Other Names: Educational intervention with eGuide to colonoscopy

SUMMARY:
The investigators will attempt to improve the patient experience before colonoscopy. The investigators will provide an in-office ipad video series and an electronic web guide to help patients learn all the best ways to prepare for colonoscopy. The investigators will then follow the patients who receive this eGuide to colonoscopy and observe whether or not they enjoyed the additional access to information from their providers, and will monitor whether or not they were better prepared for their colonoscopy.

DETAILED DESCRIPTION:
This study would assess the ability of an e-intervention in patient education and instructions during peri-procedure and procedural day visits to improve the experience of gastroenterology procedures. This study would seek to show that through this alternative educational measure, there would be an increased show rate to colonoscopy appointments, an increased preparation quality, and an increase in patient understanding and satisfaction with the colonoscopy procedure. The investigators will attempt to track procedure completion rate and polyp detection rate for individual providers.

The e-intervention would be multimodal. In the pre-procedure setting, ipad would be able to provide a viewpoint for the video education, a template for the patients (or caregivers) to send themselves links to appropriate instructions to remind them of their obligations by secure email. This e-intervention would supplement traditional printed and website accessible instructions.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Colonoscopy at Johns Hopkins
* Ages 18 to 90
* Access to email (themselves or designee)
* Access to internet outside of physician visit

Exclusion Criteria:

* Unable to consent
* Unwilling to participate
* Unable to care for themselves

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Completion rate of colonoscopy procedure | 1 day
  Could the colonoscopy be completed in its entirety on the date scheduled?

SECONDARY OUTCOMES:
preparation quality | one day
  What was the quality of preparation as measured on the day of colonoscopy, preferably by the Boston Bowel Preparation score.
adenoma detection rate by provider | 6 months
  Measurement of adenoma detection rate by provider for study patients.
Patient satisfaction | 3 months
  An individual patient satisfaction survey will be provided to patients via the eGuide to Colonoscopy web-portal and will assess their enjoyment and understanding. A patient satisfaction survey is employed by the division to random patients over a three month period. We will assess both of these to determine patient satisfaction with the study intervention.

OTHER OUTCOMES:
Feasibility of intervention in practice | 1 year
  What is the feasibility of the intervention? Could providers and patients navigate the eGuide? Was theft a problem with having Ipads in the office space? Was the home webportal of the eGuide able to be accessed by patients receiving information in the office?

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Stein, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States